CLINICAL TRIAL: NCT04519684
Title: A Phase IB/IIA Study of Allogeneic Bone Marrow Derived Mesenchymal Stem Cells for the Treatment of Ileal Anal Anastomosis and Ileal Pouch Fistulas in the Setting of Crohn's Disease of the Pouch
Brief Title: Study of Mesenchymal Stem Cells for the Treatment of Ileal Pouch Fistula's in Participants With Crohn's Disease
Acronym: IPAAF
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amy Lightner (Other)
Responsible Party: Sponsor-Investigator, Amy Lightner, Sponsor-investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20-818
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Ileal Pouch; Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cells (Experimental): Direct injection of allogeneic bone marrow derived mesenchymal stem cells at a dose of 75 million cells into the ileal pouch fistula(s) at baseline with a possible repeat injection at 3 months if not completely healed from the first injection.
  Interventions: Drug: Mesenchymal stem cells
- Placebo (Placebo Comparator): Direct injection of normal saline. If not completely healed after 6 months, participants will then cross over to the treatment group to receive a direct injection of allogeneic bone marrow derived mesenchymal stem cells at a dose of 75 million cells into ileal pouch fistula(s).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mesenchymal stem cells — Allogeneic bone marrow derived mesenchymal stem cells
  Arms: Mesenchymal stem cells
Other: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
Restorative proctocolectomy with ileal pouch anal anastomosis (IPAA) is the procedure of choice for patients with ulcerative colitis, familial adenomatous polyposis, and select patients with Crohn's disease due to overall low patient morbidity and good quality of life. However, some patients can develop Crohn's disease of the pouch, a clinical diagnosis of Crohn's disease following IPAA. One of the manifestations of Crohn's disease of the pouch includes a fistula from the pouch that travels to the vagina or perianal area. These fistulas can be quite difficult to manage with medications and local surgical intervention, and, on occasion result in a reconstruction pouch but more often require a pouch excision with permanent end ileostomy. The purpose of this study is to evaluate the safety and efficacy of using allogeneic bone marrow derived mesenchymal stem cells to treat people who have a peri-pouch fistula related to a clinical diagnosis of Crohn's disease of the pouch.

DETAILED DESCRIPTION:
This aim of this study is to determine the safety and efficacy of adult allogeneic bone marrow derived mesenchymal stem cells (MSCs), for the treatment of medically refractory peri-pouch fistulizing disease in the setting of Crohn's disease of the pouch. The study will randomize 20 participants. Enrolled participants will be randomized to treatment group with MSCs, versus placebo in a 3:1 fashion. Participants in the treatment group will have a direct injection of MSCs at a dose of 75 million cells. This will be given as a direct injection in and around the fistula tract. Participants will be evaluated for complete healing at three months. If complete healing has been achieved participants will continue to be followed for one year. If complete healing has not been achieved at three months, participants will be eligible for a second injection of MSCs at the same dose of 75 million cells. Control participants without complete healing from placebo will cross over at the 6 month visit to receive an injection of MSCs and will be followed for one year after treatment to a total duration of 18 months. The primary efficacy analysis will be conducted at the month 6 time point.

ELIGIBILITY:
Inclusion Criteria

1. Men and women 18-75 years of age who have undergone an ileal pouch anal anastomosis at least 6 months prior who have developed a clinical diagnosis of Crohn's disease of the pouch as determined by a combination of clinical symptoms, pouchoscopy with biopsy, enterography.
2. Single and multi-tract (up to 2 internal and 3 external openings) fistula tract arising from the ileal pouch, ileal anal anastomosis, or anal canal distal to anastomosis that travels to the perianal skin, perineal body, or vagina. Patients with fistulas that arise from the pouch, anastomosis, or anal canal distal to the anastomosis will both be included in enrollment.

   1. Acceptable internal openings and tract locations for the fistula to arise from include the ileal pouch body, the pouch anal anastomosis, and the anal canal distal to the anastomosis.
   2. Acceptable external openings and tract locations for the fistula to arise from include the perianal skin, perineal body, and/or the vaginal wall.
3. Concurrent Crohn's related therapies with stable doses (>2 months) corticosteroids, 5-ASA drugs, immunomodulators, anti-TNF therapy, anti-integrin and anti-interleukin are permitted.
4. Have failed conventional medical therapies described above, defined as a lack of response to systemic immune suppression (e.g. azathioprine, methotrexate, 6-mercaptopurine) or biologic (e.g. anti-TNF, anti-integrin, anti-interleukin) therapies to treat fistulizing CD for at least 2 months
5. Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
6. Competent and able to provide written informed consent
7. Ability to comply with protocol.

Exclusion Criteria

1. Inability to give informed consent.
2. Severe antibiotic refractory pouchitis
3. Severe cuffitis refractory to antibiotics
4. Change in medical management for CD in the previous 2 months or changes anticipated in the next 2 months
5. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the subject.
6. Specific exclusions;

   1. HIV
   2. Hepatitis B or C
   3. Abnormal CBC at screening

   i. Platelets <50 kg/uL or greater than 1.5 million kg/uL ii. WBC <50 x kg/uL iii. Hbg <7.0 g/dL d. Abnormal AST or ALT at screening(defined as >/= 2x ULN)
7. History of cancer including melanoma (with the exception of localized skin cancers) within one year of screening
8. History of colorectal cancer within 5 years
9. Investigational drug within thirty (30) days of baseline
10. Pregnant or breast feeding or trying to become pregnant
11. Branching fistula tract that has > 2 internal openings or 3 external openings,

    1. Subjects with greater than 3 blind/branching tracts are excluded
    2. Fistula tracts on the left and/or right side are allowed
12. Allergic to local anesthetics
13. Unwilling to agree to use acceptable contraception methods during participation in study
14. Subjects with a non-abscessed chronic cavity will not be included in enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events | Month 6
  Number of participants with treatment related adverse events post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease as assessed by protocol CCF-Stem Cells IBD-002

SECONDARY OUTCOMES:
Complete clinical healing | Month 6, Month 12
  Number of participants with complete clinical healing post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease of the pouch.
  Complete Healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 3 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical Healing: 100% cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
Partial healing | Month 6, Month 12
  Number of participants with partial clinical healing,post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease
  Partial Healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 2 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical healing: Greater than or equal to 50 % cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
Lack of response | Month 6, Month 12
  Number of participants with lack of response post-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease
  Lack of Response is defined as: Radiographic and Clinical healing which does not meet the threshold for Partial Healing
Worsening disease | Month 6, Month 12
  Number of participants with worsening disease-injection of 75 million allogeneic bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease
  Worsening Disease is defined as:
  Radiographic: MRI with a fluid collection >2 cm in 2 of 3 dimensions, edema, inflammation or sign of active inflammatory response. An increased number of tracts may be seen, or increased branching from the primary tract,
  Clinical: Increased drainage per patient report and on clinical exam

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lightner, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fazio VW, Kiran RP, Remzi FH, Coffey JC, Heneghan HM, Kirat HT, Manilich E, Shen B, Martin ST. Ileal pouch anal anastomosis: analysis of outcome and quality of life in 3707 patients. Ann Surg. 2013 Apr;257(4):679-85. doi: 10.1097/SLA.0b013e31827d99a2. PMID 23299522
- [Background] Ozdemir Y, Kiran RP, Erem HH, Aytac E, Gorgun E, Magnuson D, Remzi FH. Functional outcomes and complications after restorative proctocolectomy and ileal pouch anal anastomosis in the pediatric population. J Am Coll Surg. 2014 Mar;218(3):328-35. doi: 10.1016/j.jamcollsurg.2013.11.019. Epub 2013 Nov 26. PMID 24468224
- [Background] Remzi FH, Fazio VW, Kirat HT, Wu JS, Lavery IC, Kiran RP. Repeat pouch surgery by the abdominal approach safely salvages failed ileal pelvic pouch. Dis Colon Rectum. 2009 Feb;52(2):198-204. doi: 10.1007/DCR.0b013e31819ad4b6. PMID 19279412
- [Background] Belliveau P, Trudel J, Vasilevsky CA, Stein B, Gordon PH. Ileoanal anastomosis with reservoirs: complications and long-term results. Can J Surg. 1999 Oct;42(5):345-52. PMID 10526518
- [Background] Foley EF, Schoetz DJ Jr, Roberts PL, Marcello PW, Murray JJ, Coller JA, Veidenheimer MC. Rediversion after ileal pouch-anal anastomosis. Causes of failures and predictors of subsequent pouch salvage. Dis Colon Rectum. 1995 Aug;38(8):793-8. doi: 10.1007/BF02049833. PMID 7634973
- [Background] Molendijk I, Bonsing BA, Roelofs H, Peeters KC, Wasser MN, Dijkstra G, van der Woude CJ, Duijvestein M, Veenendaal RA, Zwaginga JJ, Verspaget HW, Fibbe WE, van der Meulen-de Jong AE, Hommes DW. Allogeneic Bone Marrow-Derived Mesenchymal Stromal Cells Promote Healing of Refractory Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2015 Oct;149(4):918-27.e6. doi: 10.1053/j.gastro.2015.06.014. Epub 2015 Jun 25. PMID 26116801
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Diez MC, Tagarro I, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Long-term Efficacy and Safety of Stem Cell Therapy (Cx601) for Complex Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2018 Apr;154(5):1334-1342.e4. doi: 10.1053/j.gastro.2017.12.020. Epub 2017 Dec 24. PMID 29277560
- [Background] Panes J, Garcia-Olmo D, Van Assche G, Colombel JF, Reinisch W, Baumgart DC, Dignass A, Nachury M, Ferrante M, Kazemi-Shirazi L, Grimaud JC, de la Portilla F, Goldin E, Richard MP, Leselbaum A, Danese S; ADMIRE CD Study Group Collaborators. Expanded allogeneic adipose-derived mesenchymal stem cells (Cx601) for complex perianal fistulas in Crohn's disease: a phase 3 randomised, double-blind controlled trial. Lancet. 2016 Sep 24;388(10051):1281-90. doi: 10.1016/S0140-6736(16)31203-X. Epub 2016 Jul 29. PMID 27477896
- [Derived] Lightner AL, Reese J, Ream J, Nachand D, Jia X, Pineiro AO, Dadgar N, Steele S, Hull T. A Phase IB/IIA Study of Allogeneic, Bone Marrow-derived, Mesenchymal Stem Cells for the Treatment of Refractory Ileal-anal Anastomosis and Peripouch Fistulas in the Setting of Crohn's Disease of the Pouch. J Crohns Colitis. 2023 Apr 19;17(4):480-488. doi: 10.1093/ecco-jcc/jjac172. PMID 36322714